CLINICAL TRIAL: NCT00184951
Title: Pharmacodynamics and Pharmacokinetics of Combined Use of Rosuvastatin (Crestor) and Lopinavir/Ritonavir (Kaletra) in HIV-infected Patients With Hyperlipidemia (ROSALKA)
Brief Title: Pharmacokinetic Study of Rosuvastatin and Lopinavir/Ritonavir in HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Abbott (Industry); AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 03.01
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; Hyperlipidemia
Keywords: HIV
MeSH Terms: conditions — HIV Infections; Hyperlipidemias | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
open-label, multiple dose, single-group, 12 week trial in HIV-infected patients with hyperlipidemia while using lopinavir/ritonavir; both male or female subjects.

DETAILED DESCRIPTION:
To determine the effect of rosuvastatin on plasma lipids, lipoproteins, and endothelial function in HIV-infected patients on stable lopinavir/ritonavir therapy and to evaluate the safety of combined use of rosuvastatin and lopinavir/ritonavir. Also to determine the effect of lopinavir/ritonavir on the pharmacokinetics of rosuvastatin compared to historical controls an to determine the effect of rosuvastatin on the pk of lopinavir/ritonavir compared to historical controls and by intrapatient comparison.

ELIGIBILITY:
Inclusion Criteria:

* use of lopinavir 400mg/ritonavir 100mg bid > 3months
* HIV-1 RNA <400cop/mL
* fasting total cholesterol > 6.2mmol/L

Exclusion Criteria:

* history of sensitivity/idiosyncrasy to the drug or compounds used
* history or current condition that might interfere with absorption,distribution metabolism or excretion
* pregnant or breast-feeding
* serum transaminase levels >3 times upper limit of normal, creatinine clearance <60ml/min
* fasting plasma triglycerides level >8.0 mmol/L
* history of statin-related rhabdomyolysis or inheritable muscle diseases in family history
* clinical symptoms of myopathy or abnormal CK level
* change in antiretroviral medication within the 3 months immediately preceding first dose of rosuvastatin
* use of any statin or fibrate within 6 weeks immediately preceding first dose of rosuvastatin
* concomitant use of medications that interfere with rosuvastatin or lopinavir pharmacokinetics
* active hepatobiliary or hepatic disease
* hypothyroidism
* alcohol abuse
* japanese or chinese patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-04; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics on week 0,4,8 and 12

SECONDARY OUTCOMES:
evaluation of lipid lowering activity on week 0,4,8,12
endothelial function will be measured at week 0 & 12 (optional for patients from Leiden and Nijmegen)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Burger, Dr, Principal Investigator — Radboud University Medical Center
Locations (5):
- Germany (2):
  - University of Bonn, Bonn
  - University of Cologne, Cologne
- Netherlands (3):
  - University of Amsterdam, Amsterdam
  - University of Leiden, Leiden
  - University of Nijmegen, Nijmegen

REFERENCES:
- [Result] van der Lee M, Sankatsing R, Schippers E, Vogel M, Fatkenheuer G, van der Ven A, Kroon F, Rockstroh J, Wyen C, Baumer A, de Groot E, Koopmans P, Stroes E, Reiss P, Burger D. Pharmacokinetics and pharmacodynamics of combined use of lopinavir/ritonavir and rosuvastatin in HIV-infected patients. Antivir Ther. 2007;12(7):1127-32. PMID 18018771